CLINICAL TRIAL: NCT04251117
Title: An Open-label, Multi-center, Phase I/IIa Study of a Personalized Neoantigen DNA Vaccine (GNOS-PV02) and Plasmid Encoded IL-12 (INO-9012) in Combination with Pembrolizumab (MK-3475) in Subjects with Advanced Hepatocellular Carcinoma
Brief Title: GNOS-PV02 Personalized Neoantigen Vaccine, INO-9012 and Pembrolizumab in Subjects with Advanced HCC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Geneos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT-30
Record Dates: First submitted 2020-01-27; First posted 2020-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: HCC
MeSH Terms: interventions — rocakinogene sifuplasmid; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- GNOS-PV02 + INO-9012 + Pembrolizumab (Experimental): First line therapy with standard of care tyrosine kinase inhibitors (TKI) during which patient-specific GNOS-PV02 will be manufactured.
  GNOS-PV02 + INO-9012 + Pembrolizumab will be administered upon disease progression or intolerance to TKI.
  Interventions: Biological: GNOS-PV02; Biological: INO-9012; Drug: Pembrolizumab; Device: CELLECTRA®2000 EP Device

INTERVENTIONS:
Biological: GNOS-PV02 — GNOS-PV02 delivered by intradermal injection and electroporation
Biological: INO-9012 — INO-9012 delivered by intradermal injection and electroporation
Drug: Pembrolizumab — Pembrolizumab administered as an intravenous (IV) infusion
Device: CELLECTRA®2000 EP Device — CELLECTRA® 2000 Device is a system indicated for use to enhance the uptake and expression of plasmid-based biologics in order to enhance vaccine efficacy.

SUMMARY:
This is a single-arm, open-label, multi-site Phase I/IIa study of a personalized neoantigen DNA vaccine (GNOS-PV02) and plasmid encoded IL-12 (INO-9012) in combination with pembrolizumab (MK-3475) in subjects with histologically or cytologically confirmed diagnosis of HCC based on pathology report.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the study. The subject may also provide consent for Future Biomedical Research (FBR). However, the subject may participate in the main study without participating in FBR.
2. 18 years of age on day of signing informed consent.
3. Have histologically or cytologically confirmed diagnosis of HCC based on pathology report. Radiological diagnosis is valid to initiate screening pending confirmation by pathology.
4. Have Barcelona Clinic Liver Cancer (BCLC) Stage C disease or BCLC Stage B disease not amenable to locoregional therapy, or refractory to locoregional therapy, and not amenable to a curative treatment approach.
5. Have a Child-Pugh Class A liver score.
6. Have a predicted life expectancy of greater than 6 months.
7. Have measurable disease based on RECIST 1.1.
8. Have a performance status of 0 or 1 using the ECOG Performance Scale within 7 days of first dose of study drug.
9. Receiving or eligible for first-line therapy with sorafenib or lenvatinib.
10. Willing to submit a tissue sample for personalized DNA vaccine manufacturing.
11. Patients with chronic or acute HBV infection [as characterized by positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibodies (anti-HBcAb) with detectable HBV DNA (≥10 IU/ml)] must be treated with effective antiviral therapy, as per institutional practices, prior to enrollment and for the duration of the study therapy. Patients who test positive for anti-hepatitis B core (HBc) with undetectable HBV DNA (<10 IU/ml) do not require anti-viral therapy prior to enrollment however these subjects will be tested at every cycle to monitor HBV DNA levels and initiate antiviral therapy if HBV DNA is detected (≥10 IU/ml). Subjects with chronic infection by hepatitis C virus (HCV), who are untreated, are allowed on study. In addition, subjects with successful HCV treatment (defined as sustained virologic response [SVR] 12 or SVR 24) are allowed, as long as 4 weeks have passed between completion of HCV therapy and start of study drug. Subjects receiving antiviral therapy during TKI may be enrolled.
12. Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test for the patient to be eligible for trial enrolment.
13. Be willing to use an adequate method of contraception for the course of the study through 150 days after the last dose of study drug (male and female subjects of childbearing potential).

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
14. Demonstrate adequate organ function

Exclusion Criteria:

1. Is currently participating and receiving study drug or has participated in a study of an investigational agent and received study drug or used an investigation device, within 4 weeks of the first dose of treatment. Subjects must also have recovered from associated therapy (i.e., to Grade ≤1 or baseline) and from AEs due to any prior therapy.
2. Has received sorafenib or lenvatinib within 14 days of first dose of study drug.
3. Has had esophageal or gastric variceal bleeding within the last 6 months. If suspected, subjects will be screened for esophageal varices. If varices are present, they should be treated according to institutional standards before starting study treatment.
4. Has clinically apparent ascites on physical examination. Note: only ascites detectable on imaging studies is allowed.
5. Evidence of portal vein invasion based on imaging is allowed pending subjects meet laboratory criteria for enrollment.
6. Has had encephalopathy in the last 6 months. Subjects on rifaximin or lactulose to control their encephalopathy are not allowed.
7. Had a solid organ or hematologic transplant.
8. Had prior systemic therapy for HCC other than sorafenib or lenvatinib.
9. Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., T4, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
11. Has received locoregional therapy to liver (transarterial chemoembolization [TACE], transarterial embolization [TAE], radiation, radioembolization, or ablation) or major surgery to liver or other site within 3 weeks prior to the first dose of study drug. Minor surgery (e.g., simple excision, tooth extraction) must have occurred at least 7 days prior to the first dose of study drug (Cycle 1, Day 1). Subjects must have recovered adequately (i.e., Grade ≤1 or baseline) from the toxicity and/or complications from any intervention prior to starting therapy.
12. Has a diagnosed additional malignancy within 5 years prior to first dose of study drug, with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or curatively resected in situ cervical and/or breast cancers. Subjects with history of early-stage prostate cancer that has been curatively treated or appropriate for observation may be enrolled.
13. Has radiographically detectable (even if asymptomatic and/or previously treated) central nervous system (CNS) metastases and/or carcinomatous meningitis, as assessed by local site investigator.
14. Has a known history of, or any evidence of, interstitial lung disease or active non- infectious pneumonitis.
15. Has an active infection requiring systemic therapy.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator, including dialysis.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
18. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 150 days after the last dose of study drug.
19. Has received prior immunotherapy including anti-programmed death (PD) 1, anti-programmed death ligand (PD-L)-1, or anti-PD-L2 agents, or personalized therapies such as adoptive cell therapy or neoantigen-based vaccine.
20. Has a known history of human immunodeficiency virus (HIV) (HIV I/II antibodies).
21. Has untreated active hepatitis B virus (HBV), unless planned antiviral therapy during TKI.

    Note: Patients with HBV infection, characterized by positive HBsAg and/or HBcAb with detectable HBV DNA (≥10 IU/ml or above the limit of detection per local lab standard), must be treated with antiviral therapy as per institutional practice to ensure adequate viral suppression (HBV DNA ≤2000 IU/mL) prior to treatment with the study drug. Patients who test positive for HBcAg with undetectable HBV DNA (<10 IU/ml or under the limit of detection per local lab standard) do not require anti-viral therapy prior to enrollment.
22. Has received a live vaccine within 30 days of planned start of study treatment (Cycle 1, Day 1).

    Note: The killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Non-live COVID-19 vaccines are allowed.
23. Any contraindication for treatment with the CELLECTRA® 2000 Device:

    Less than two acceptable sites available for ID injection and EP considering the deltoid and anterolateral quadriceps muscles:
    1. Tattoos, keloids or hypertrophic scars located within 2 cm of intended administration site.
    2. Implantable-Cardioverter-defibrillator (ICD) or pacemaker (to prevent a life-threatening arrhythmia) that is located ipsilateral to the deltoid injection site (unless deemed acceptable by a cardiologist).
    3. Any metal implants or implantable medical device within the intended treatment site (i.e. electroporation area).
24. Has no mutations detected after sequencing of the tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2028-11-29 (Estimated)

PRIMARY OUTCOMES:
Adverse evets as graded by CTCAE v5.0 | Up to 24 Months
Immunogenicity of a personalized neoantigen DNA vaccine as measured by interferon-γ secreting T lymphocytes in peripheral blood mononuclear cells (PBMCs) using ELISpot | Up to 24 Months
Immunogenicity of a personalized neoantigen DNA vaccine as measured by T-cell activation and cytolytic cell phenotype in PBMCs using Flow Cytometry | Up to 24 Months

SECONDARY OUTCOMES:
Anti-tumor activity as measured by Objective Response Rate (ORR) by RECIST 1.1 by investigator review | Up to 24 Months
Anti-tumor activity as measured by ORR by iRECIST | Up to 24 Months
Anti-tumor activity as measured by Duration of Response (DOR) | Up to 24 Months
Anti-tumor activity as measured by Disease Control Rate (DCR) | Up to 24 Months
Anti-tumor activity as measured by Progression Free Survival (PFS) as assessed by RECIST 1.1 | Up to 24 Months
Anti-tumor activity as measured by Progression Free Survival (PFS) as assessed by iRECIST | Up to 24 Months
Anti-tumor activity as measured by Overall Survival (OS) | Up to 24 Months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
- Auckland Clinical Studies, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yarchoan M, Gane EJ, Marron TU, Perales-Linares R, Yan J, Cooch N, Shu DH, Fertig EJ, Kagohara LT, Bartha G, Northcott J, Lyle J, Rochestie S, Peters J, Connor JT, Jaffee EM, Csiki I, Weiner DB, Perales-Puchalt A, Sardesai NY. Personalized neoantigen vaccine and pembrolizumab in advanced hepatocellular carcinoma: a phase 1/2 trial. Nat Med. 2024 Apr;30(4):1044-1053. doi: 10.1038/s41591-024-02894-y. Epub 2024 Apr 7. PMID 38584166
- See also: Nature Medicine — https://www.nature.com/articles/s41591-024-02894-y